CLINICAL TRIAL: NCT04519931
Title: The Effect of Using a Stress Ball on Pain, Anxiety and Satisfaction During the Endoscopy Procedure
Brief Title: The Effect of Stress Ball Used During Endoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi (Other)
Responsible Party: Principal Investigator, Elif Gezginci, Rn, PhD, Asst Prof., Saglik Bilimleri Universitesi
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20-85
Record Dates: First submitted 2020-08-17; First posted 2020-08-20 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Pain; Anxiety; Satisfaction
Keywords: anxiety; endoscopy; pain; nursing; stress ball
MeSH Terms: conditions — Pain; Anxiety Disorders; Personal Satisfaction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Stress ball (Experimental)
  Interventions: Other: Stress ball
- Control group (No Intervention)

INTERVENTIONS:
Other: Stress ball — The stress ball is a toy, usually no larger than 7 cm. It is used to relieve stress and muscle tension. Stress ball is one of the cognitive and behavioral therapy methods used in pain control. Stress ball is used as a method of diverting attention during painful procedures. It appears to reduce pain and anxiety.
  Arms: Stress ball

SUMMARY:
Endoscopy procedure is a frequently used method in the evaluation of the gastrointestinal system. Upper gastrointestinal system endoscopy can be performed with and without sedation. Sedation is the controlled sleep of the patient with certain drugs (pharmacological methods). Non-pharmacological methods help reduce anxiety and pain. In this study, a non-pharmacological stress ball will be used. It is aimed to evaluate the effect of using a stress ball on pain, anxiety and satisfaction during upper gastrointestinal system endoscopy.

DETAILED DESCRIPTION:
Patients do not want to think that an upper GIS endoscopy without sedation will be difficult. However, some complications can be seen like hypoxemia, allergic reaction, malignant hyperthermia, hypoventilation, respiratory depression, hypotension, bradycardia, apnea, hypoxia, etc. due to sedation applied during endoscopy.

Non-pharmacological methods help reduce anxiety and pain. Although sedative and analgesic medications reduce anxiety and relieve pain, endoscopy is still painful for patients. During the endoscopy process, non-pharmacological methods are used to draw attention to another direction, but it is not encountered that the stress ball is used as one of these methods in the endoscopy procedure.

This study was planned as a single-center prospective randomized controlled study for the treatment of the stress ball method used during the endoscopy procedure, pain in anxiety and satisfaction levels.

The data obtained in the study will be analyzed using the SPSS (Statistical Package for Social Sciences) for Windows 22.0 program. Number, percentage, mean, standard deviation will be used as descriptive statistical methods in the evaluation of data. In comparing the difference between two independent groups, Student's t test will be used for data conforming to normal distribution, and Mann-Whitney U test will be used for data that do not comply with normal distribution. The difference between two repeated measurements will be analyzed with dependent groups t-test for data conforming to normal distribution, and Wilcoxon test for data that do not conform to normal distribution. The difference between three and more measurements that do not comply with the normal distribution will be compared with the analysis of variance in repeated measures for data that do not fit the normal distribution, and with the Friedman test for data that do not comply with the normal distribution. A value of P <0.05 will be considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* To have an upper gastrointestinal endoscopy for the first time
* Not wanting sedation during upper gastrointestinal endoscopy
* Being between the ages of 18-75
* Being willing to participate in research

Exclusion Criteria:

* Using analgesic or anesthetic drugs before or during the procedure
* Using antidepressants, anxiolytic and sedative drugs
* Having communication difficulties and mental disability

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2020-11-05 (Actual); Primary Completion 2021-03-04 (Actual); Study Completion 2021-09-01 (Actual)

PRIMARY OUTCOMES:
Change on pain intensity as measured by Visual Analog Scale | just before procedure, during, and just after procedure
  The average score change on pain intensity as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure pain intensity. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that pain intensity is high.

SECONDARY OUTCOMES:
Score change on anxiety level as measured by State-Trait Anxiety Inventory | just before and after procedure
  The average score change on anxiety level as measured by State-Trait Anxiety Inventory. This scale in used to measure anxiety. The scores on the scale ranges from 20 to 80. The high scores on the scale indicate that anxiety is high.

OTHER OUTCOMES:
Change on satisfaction level as measured by Visual Analog Scale | just after procedure
  The average score change on satisfaction level as measured by Visual Analog Scale. This scale is an unidimensional measure commonly used to measure satisfaction level. The scale is a measuring tool with length of 0-10 cm. High scores on the scale indicate that satisfaction level is high.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Gezginci, RN, PhD, Principal Investigator — Saglik Bilimleri Universitesi
Locations (1):
- University of Health Sciences Turkey, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Karatas TC, Gezginci E. The Effect of Using a Stress Ball During Endoscopy on Pain, Anxiety, and Satisfaction: A Randomized Controlled Trial. Gastroenterol Nurs. 2023 Jul-Aug 01;46(4):309-317. doi: 10.1097/SGA.0000000000000739. Epub 2023 May 17. PMID 37199436